CLINICAL TRIAL: NCT01992237
Title: Pilot Study of Measuring Energy Expenditure in ECMO Patients Under Consideration of Type of Ventilation and to Approximate Cardiac Output
Brief Title: Measuring Energy Expenditure in ECMO (Extracorporeal Membrane Oxygenation) Patients
Acronym: MEEP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Steffen Weber-Carstens, PD Dr. med. Steffen Weber-Carstens, Charite University, Berlin, Germany
Other Study IDs: Charité-MEEP-01
Record Dates: First submitted 2013-10-21; First posted 2013-11-25 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Acute Lung Injury; Respiratory Distress Syndrome, Adult
Keywords: ALI,; ARDS,; ECMO,; energy expenditure,; mechanical ventilation,; Extracorporeal Membrane Oxygenation; Nutrition Assessment; Pulmonary Ventilation
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood will be obtained for metabolomic analyses.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ALI patients: Patients with ARDS by Berlin definition and with or without clinical indication for ECMO treatment.

SUMMARY:
With the perception that lung protective ventilation with regard to low tidal volume ventilation and limiting airway pressures improves outcome in ARDS (acute respiratory distress syndrome) and that the development of new technical devices of extracorporeal lung assist systems with lower complication rates support establishment of lung protective ventilation strategies these systems are more and more frequently used. All critically ill patients with and without ECLA (extracorporeal lung assist)/ECMO (extracorporeal membrane oxygenation) treatment are on high risk for muscle wasting, leading to more comorbidity and higher mortality risk. Besides inflammation malnutrition is known as one of the main risk factors. Over and underfeeding should be prevented. However nutritional aspects of patients on extracorporeal lung assist are hardly investigated. Up to now changes in metabolic rates induced by ECLA/ECMO are poorly described. Factors like work of breathing, changes in cardiac output and septic state are influencing energy metabolism but until now there is no tool for measuring energy expenditure in clinical routine for patients on ECLA/ECMO. Indirect calorimetry is a simple device only for patients without ECLA/ECMO system. Oxygenation and CO2 (carbon dioxide) elimination by the lung assist system can be calculated but is not implemented to clinical routine. The combination of indirect calorimetry and calculation of lung assist function at the same time would give us the chance to adapt nutrition rates to energy expenditure. This may prevent muscle wasting and weakness. This pilot study will include 40 participating patients during 8 month investigating nutritional therapy adapted to energy expenditure calculated by O2 and CO2 turnover rates in patients on ECLA or ECMO systems. The investigators aim is to describe a calculation to set nutrition targets in ECMO patients. Second the investigators will describe level of nutritional needs under consideration of different mechanical ventilation states. Third O2 consumption and CO2 elimination will be used to estimate cardiac output.

ELIGIBILITY:
Inclusion Criteria:

* critically ill patients with ALI
* informed consent by the patients or legal proxy

Exclusion Criteria:

* age < 18
* no informed consent by the patients or legal proxy
* pregnancy
* infaust prognosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ALI
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-10; Primary Completion 2018-01 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Energy expenditure in kcal | Once within first week after ICU admission for 20 minutes
  Measurement of energy expenditure before ECMO use.
Energy expenditure in kcal | Once within first week after ECMO /ECLA treatment started for 20 minutes
  Measurement and calculation of energy expenditure with ECMO / ECLA use and controlled mechanical ventilation.
Energy expenditure in kcal | Once within first week after ECMO /ECLA was removed for 20 minutes
  Measurement of energy expenditure with ECMO / ECLA use.

SECONDARY OUTCOMES:
Energy expenditure in kcal | Once during ECMO / ECLA treatment and controlled mechanical ventilation for 20 minutes
  Measuring and calculating energy expenditure under consideration of ventilation support for controlled pressure ventilation.
Energy expenditure in kcal | Once during ECMO / ECLA treatment and spontaneous breathing with supportive mechanical ventilation for 20 minutes
  Measuring and calculating energy expenditure under consideration of ventilation support. Spontaneous breathing with supportive mechanical ventilation and during ECMO / ECLA treatment.
Energy expenditure in kcal | Once during ECMO / ECLA treatment and spontaneous breathing with supportive mechanical ventilation for 20 minutes
  Measuring and calculating energy expenditure under consideration of ECMO /ECLA treatment it self. Spontaneous breathing with supportive mechanical ventilation and during ECMO / ECLA treatment without gas flow just before ECMO / ECLA removal.
Estimation of cardiac output in liter per minute | Calculated from the six measurements of the energy expenditure (as described above) during the ICU stay
  Approximately calculation of cardiac output by O2 and CO2 metabolism and compared to cardiac output measurements by cardiac echo and measurements of thermodilution.

OTHER OUTCOMES:
Comparing cardiac parameters measured by echo with parameters calculated by right heart catheter | Calculated from the six measurements of the energy expenditure (as described above) an clinical routine measurements during the ICU stay
  If patients get a right heart catheter by clinical reason and echo investigations we will compare these values for equal time-points.

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Weber-Carstens, MD, Principal Investigator — Charité - Universitätsmedizin Berlin, Department of Anesthesiology and Intensive Care Medicine
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Result] Wollersheim T, Frank S, Muller MC, Skrypnikov V, Carbon NM, Pickerodt PA, Spies C, Mai K, Spranger J, Weber-Carstens S. Measuring Energy Expenditure in extracorporeal lung support Patients (MEEP) - Protocol, feasibility and pilot trial. Clin Nutr. 2018 Feb;37(1):301-307. doi: 10.1016/j.clnu.2017.01.001. Epub 2017 Jan 16. PMID 28143666
- [Derived] Muller MC, Wilke SK, Dobbermann A, Kirsten S, Russ M, Weber-Carstens S, Wollersheim T. Dissolved Oxygen Relevantly Contributes to Systemic Oxygenation During Venovenous Extracorporeal Membrane Oxygenation Support. ASAIO J. 2024 Aug 1;70(8):667-674. doi: 10.1097/MAT.0000000000002171. Epub 2024 Mar 6. PMID 38446867
- [Derived] Muller MC, Wilke SK, Dobbermann A, Carbon NM, Lammel S, Russ M, Weber-Carstens S, Wollersheim T. Quantitative Gas Exchange in Extracorporeal Membrane Oxygenation-A New Device: Accuracy, Approach-based Difficulties, and Caloric Targeting. ASAIO J. 2023 Jan 1;69(1):61-68. doi: 10.1097/MAT.0000000000001662. Epub 2022 Jan 31. PMID 35759721